CLINICAL TRIAL: NCT02077868
Title: Evaluation of an Immunomodulatory Maintenance Treatment in Patients With Metastatic Colorectal Cancer With Tumor Reduction During Induction Treatment
Brief Title: Evaluation of MGN1703 Maintenance Treatment in Patients With mCRC With Tumor Reduction During Induction Treatment
Acronym: IMPALA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mologen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGN1703-C06
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: CRC; mCRC; maintenance treatment; immune modulation; colorectal cancer; immunotherapy; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm A (Other): Patients in Control Arm A receive usual maintenance Treatment according to local investigator's decsision
  Interventions: Other: Usual Maintenance
- Treatment Arm B (Experimental): MGN1703 treatment as maintenance therapy
  Interventions: Drug: MGN1703 treatment

INTERVENTIONS:
Other: Usual Maintenance — Usual maintenance therapy according to local investigator's practice, e.g. treatment break, reduced treatment, continued treatment, and other
  Arms: Control Arm A
Drug: MGN1703 treatment — MGN1703 will be used as single agent maintenance treatment
  Other Names: dSLIM
  Arms: Treatment Arm B

SUMMARY:
The purpose of this this trial is to prove the efficacy and safety of MGN1703 as a maintenance therapy after first-line chemotherapeutic treatment of metastatic colorectal cancer.

DETAILED DESCRIPTION:
Due to the toxicity of chemotherapeutic medications treatment breaks are common practice in the treatment of metastatic colorectal cancer. During these treatment breaks a variety of maintenance treatments are available.

MGN1703 is developed not only to help the Patient to recover from chemotherapy but also to boost the patient's immune System and thus help him to effectively fight the Tumor himself.

After the concept has already been proved in a previous study this Trial is conducted to further evaluate the safety and efficacy of MGN1703 Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female patient 18 years or older
* Histologically confirmed diagnosis of colorectal cancer presenting with unresectable stage IV (UICC) disease (primary tumor may be present)
* Complete or partial response, as assessed by local investigators according to RECIST 1.1, within 12-30 weeks from start of induction treatment with standard first-line chemotherapy with or without biological agents
* ECOG PS 0-1
* Haematology and biochemistry laboratory results within the limits normally expected for the patient population recovering after receiving induction treatment
* Male and female patients of childbearing potential (i.e. did not undergo surgical sterilization - hysterectomy, bilateral tubal ligation, or bilateral oophorectomy - and are not post-menopausal for at least 24 consecutive months) must use an effective method of contraception. Females of child bearing potential must have a negative serum pregnancy test

Exclusion Criteria:

* History of other malignant tumors within the last 5 years, except basal cell carcinoma or curatively excised cervical carcinoma in situ
* Known brain metastases (present or treated)
* Contraindication to receiving MGN1703 as per current investigator brochure
* Known hypersensitivity to any component of the study product
* Prior allogeneic stem cell transplantation or organ transplantation
* Active or uncontrolled infections or undiagnosed febrile condition
* Severe anemia requiring repeated blood cell transfusion
* Pre-existing autoimmune or antibody-mediated diseases or immune deficiency
* Chronic systemic immune therapy or immunosuppressant medication other than steroids within the last 6 weeks; continuous systemic steroid treatment within the last 2 weeks prior to start of study treatment
* Use of systemic antibiotic therapy within the last 2 weeks prior to start of study treatment
* Inadequate pulmonary function according to the Investigator's judgment, history of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* HIV seropositivity or active HBV/HCV infection
* Serious concomitant disease or medical condition that in the judgment of the investigator renders the patient at high risk of treatment complications
* Female patient who is pregnant or breast feeding
* Contraindication to receive the planned standard maintenance treatment according to applicable SmPC
* Treatment with any anti-cancer investigational drug within 12 months prior to study treatment or participation in another clinical study with other investigational drugs within 28 days prior to study treatment
* Vaccination within 1 months prior to start of study treatment
* Any medical, mental, psychological or psychiatric condition that in the opinion of the investigator would not permit the patient to complete the study or understand the patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 36 months
  Overall survival after randomization

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 36 months
  PFS1: from randomization until first PD PFS2: from start of re-introduction therapy until second PD PFS3: from start of first-line Treatment until second PD
Safety | 36 months
  AEs, vital signs, ECGs, safety labs as required
Overall Response rate | 36 months
  Complete and partial responses according RECIST 1.1 after randomization
Quality of life (QoL) | 36 months
  QoL according EORTC questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD, Principal Investigator — Royal Marsden Hospital London
Locations (124):
- Austria (4):
  - Landesklinikum Krems, Krems
  - Kaiser-Franz-Josef-Spital, Vienna
  - Krankenhaus Hietzing, Vienna
  - Universitätsklinik Wien, Vienna
- Belgium (3):
  - Onze-Lieve-Vrouwziekenhuis VZW (OLV), Aalst
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
- Estonia (3):
  - East-Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre, Tallinn
  - University clinic Tartu, Tartu
- France (21):
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - CHRU Brest - Hôpital Morvan, Brest
  - Hôpital Henri Mondor, Créteil
  - Polyclinique du Bois, La Chaussée-Saint-Victor
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - CHU Hôpital de la Timone, Marseille
  - Centre Hospitalier Belfort-Montbéliard, Montbéliard
  - Hôpital Antoine-Béclère, Paris
  - Groupe Hosptalier Paris Saint Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou (HEGP), Paris
  - Hopital Pitie-Salpetriere, Paris
  - Gustave Roussy Cancer Campus, Paris
  - CHU de Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Clinique Saint Anne, Strasbourg Oncologie Liberale, Strasbourg
  - Hôpital Rangueil, Toulouse
- Germany (57):
  - Klinikum Augsburg, Augsburg
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Internistische Schwerpunktpraxis, Bad Reichenhall
  - Klinikum Mittelbaden Baden-Baden Balg, Baden-Baden
  - Klinikum Mittelbaden Medizinische Klinik II, Baden-Baden
  - Klinikum Bayreuth GmbH, Bayreuth
  - Charité - Universitätsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Medizinisches Versorgungszentrum Ärzteforum Seestrasse, Berlin
  - Ärzteforum Hennigsdorf, Berlin
  - St. Josef-Hospital im Katholischen Klinikum Bochum, Bochum
  - Onkologie / Hämatologie, Bottrop
  - Überörtliche Gemeinschaftspraxis, Bottrop
  - DIAKO Ev. Diakonie-Krankenhaus gemeinnützige GmbH, Bremen
  - Universitätsklinikum Köln, Cologne
  - Gefos Dortmund MBM, Dortmund
  - Onkozentrum Dresden/Freiberg, Dresden
  - Unversitätsklinikum Carl Gustav Carus, Dresden
  - Kliniken Essen-Mitte, Essen
  - Frankfurter Diakonie Kliniken, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Klinik für Tumorbiologie, Freiburg im Breisgau
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinisches Versorgungszentrum Osthessen GmbH, Fulda
  - Universitätsklinikum Gießen und Marburg, Standort Gießen, Giessen
  - MVZ Onkologische Kooperation Harz, Goslar
  - Onkologische Schwerpunktpraxis, Gütersloh
  - Universitätsklinikum Halle (Saale), Halle
  - Facharztzentrum Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Onkologische Schwerpunktpraxis Leer-Emden, Leer
  - Klinikum Leverkusen, Leverkusen
  - Onkologie Dreiländerdreieck, Loerrach
  - Onkologie Dreiländereck - Onkologische Schwerpunktpraxis Lörrach, Loerrach
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitaetsmedizin der Johannes-Gutenberg-Universitaet, Mainz
  - Klinikum Mannheim GmbH, Mannheim
  - University Hospital Marburg, Marburg
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinikum Bogenhausen, München
  - Klinikum Neuperlach, München
  - Klinikum rechts der Isar, München
  - Klinikum Nürnberg, Nuremberg
  - Pius-Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - Sana Kliniken Ostholstein, Oldenburg
  - Paracelsus-Krankenhaus Ruit, Ostfildern
  - St. Vincenz-Krankenhaus, Paderborn
  - Oncologianova GmbH, Recklinghausen
  - Elblandkliniken, Riesa
  - Vivantes Klinikum, Spandau
  - Klinikum Stuttgart - Katharinenhospital, Stuttgard
  - Kliniken Südostbayern, Traunstein
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Horst Schmidt Klinik, Wiesbaden
  - Marienhospital, Witten
  - HELIOS Klinikum Wuppertal Medizinische Klinik I, Wuppertal
- Italy (9):
  - Candiolo Cancer Institute, Candiolo
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - University Hospital San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Istituto Oncologico Veneto, Padua
  - Policlinico San Mateo, Pavia
  - Ospedale Infermi di Rimini, U.O. Oncologia, Rimini
  - Ospedale Civile SS Annunziata, U.O.C. Oncologia Medica, Sassari
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine
- Spain (20):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Parc Tauli Sabadell Hospital, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital de la Santa Creu i Sant Pau, L'Hospitalet de Llobregat
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario 12 de Octubre, Santander
  - Complejo Hospitalario Universitario, Santiago de Compostela
  - Consorcio Hospital General de Valencia, Valencia
- United Kingdom (7):
  - Aberdeen Royal Infirmary, Aberdeen
  - The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust - Royal Bournemouth Hospital, Bournemouth
  - Royal Marsden Hospital, London
  - The Christie Clinic, Manchester
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford
  - Royal Marsden Hospital, Sutton
  - York Teaching Hospitals NHS Fondation Trust, Research and Development department, York